CLINICAL TRIAL: NCT00650884
Title: Plantar Fasciopathy Treated With Dynamic Splinting: A Randomized, Controlled, Cross-Over Study
Brief Title: Plantar Fasciitis Treated With Dynamic Splinting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dynasplint Systems, Inc. (Industry)
Responsible Party: Buck Willis, PhD: Clinical Research Director, Dynasplint Systems, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Dynasplint, DYN1-08-022
Record Dates: First submitted 2008-03-31; First posted 2008-04-02 (Estimated); Last update posted 2012-04-30 (Estimated); Status verified 2012-04

CONDITIONS: Plantar Fasciitis
Keywords: Dynamic Splinting for low-load, prolonged-duration stretch
MeSH Terms: conditions — Fasciitis, Plantar | interventions — Cross-Over Studies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (No Intervention): ALL PATIENTS WILL BE TREATED WITH STANDARD OF CARE (Orthoses, NSAIDs, Home therapy instructions). CONTROL PATIENTS will only be treated with Standard of Care during this 12 week trial, but will also be treated with the Ankle Dorsiflexion Dynasplint System which delivers a low-load, prolonged-duration stretch after completion of this study.
  Interventions: Device: Ankle Dorsiflexion Dynasplint System
- 2 (Experimental): ALL PATIENTS WILL BE TREATED WITH STANDARD OF CARE (Orthoses, NSAIDs, Home therapy instructions). EXPERIMENTAL PATIENTS will also be treated with the Ankle Dorsiflexion Dynasplint System which delivers a low-load, prolonged-duration stretch while sleeping.
  Interventions: Device: Ankle Dorsiflexion Dynasplint System
- 3 (Other): ALL PATIENTS WILL BE TREATED WITH STANDARD OF CARE (Orthoses, NSAIDs, Home therapy instructions). CROSS-OVER patients will be initially treated only with Standard of Care, and after six weeks, they will be Crossed-Over and fit with the Ankle Dorsiflexion Dynasplint System which delivers a low-load, prolonged-duration stretch while sleeping.
  Interventions: Device: Ankle Dorsiflexion Dynasplint System

INTERVENTIONS:
Device: Ankle Dorsiflexion Dynasplint System — Dynamic Splinting utilizes the protocols of Low-Load, Prolonged-Duration Stretch (LLPS) with calibrated, adjustable tension to increase the Total End Range Time (TERT) to reduce contracture. This unit is worn at night while sleeping (6-8 hours) and, this does not affect activities of daily living.
  Other Names: Cross-Over

SUMMARY:
The purpose of this study is to determine if the Ankle Dorsiflexion Dynasplint System (DS) is effective in reducing pain from Plantar Fasciitis (Fasciopathy).

DETAILED DESCRIPTION:
To determine the efficacy of Ankle Dorsiflexion Dynasplint System (DS) in treating patients with plantar fasciopathy, in a multi-centered, randomized, controlled, cross-over study.

ELIGIBILITY:
Inclusion Criteria:

Patients enrolled will have been DIAGNOSED with Plantar Fasciitis which is associated with significant pain and includes the following:

* Pain on the bottom of the heel
* Pain that is usually worse upon arising or after long periods of non weight bearing
* Pain that increases over a period of months
* Pain is worsened by walking barefoot on hard surfaces or by walking up stairs
* Morning mobility limitations
* Preference of patients to "walk on their toes"
* Paresthesias after non weight bearing (while sitting or lying down or both)
* Nocturnal pain
* Patients must be willing and able to sign the informed consent

Exclusion Criteria:

* Achilles tendon injury
* Acute traumatic rupture of the plantar fascia
* Calcaneal bursitis
* Calcaneal neuritis
* Calcaneal stress fracture
* Lumbosacral radiculopathy of S1 nerve root
* Retrocalcaneal bursitis
* Tarsal tunnel syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2008-02; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Change in Foot Ankle Pain Disability Survey scores | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dr Mathew M John, DPM, Study Chair — Ankle & Foot Centers, PC; Buck Willis, PhD, Study Director — Dynasplint Systems, Inc.
Locations (4):
- United States (4):
  - Kaiser Permanente, Sacramento, California
  - Orlando Foot & Ankle Center, Orlando, Florida
  - Ankle & Foot Centers, PC, Marietta, Georgia
  - Lopez Foot Ankle Clinic, Fort Worth, Texas

REFERENCES:
- [Background] Guldemond NA, Leffers P, Sanders AP, Emmen H, Schaper NC, Walenkamp GH. Casting methods and plantar pressure: effects of custom-made foot orthoses on dynamic plantar pressure distribution. J Am Podiatr Med Assoc. 2006 Jan-Feb;96(1):9-18. doi: 10.7547/0960009. PMID 16415278
- [Background] Riddle DL, Pulisic M, Pidcoe P, Johnson RE. Risk factors for Plantar fasciitis: a matched case-control study. J Bone Joint Surg Am. 2003 May;85(5):872-7. doi: 10.2106/00004623-200305000-00015. PMID 12728038
- [Background] Riddle DL, Schappert SM. Volume of ambulatory care visits and patterns of care for patients diagnosed with plantar fasciitis: a national study of medical doctors. Foot Ankle Int. 2004 May;25(5):303-10. doi: 10.1177/107110070402500505. PMID 15134610
- [Background] Dmitri Luke BS. Plantar fasciitis: a new experimental approach to treatment. Med Hypotheses. 2002 Jul;59(1):95-7. doi: 10.1016/s0306-9877(02)00120-2. PMID 12160690
- [Background] Ross M. Use of the tissue stress model as a paradigm for developing an examination and management plan for a patient with plantar fasciitis. J Am Podiatr Med Assoc. 2002 Oct;92(9):499-506. doi: 10.7547/87507315-92-9-499. PMID 12381799
- [Background] MacKay-Lyons M. Low-load, prolonged stretch in treatment of elbow flexion contractures secondary to head trauma: a case report. Phys Ther. 1989 Apr;69(4):292-6. doi: 10.1093/ptj/69.4.292. PMID 2928396
- [Background] Willis B, John M. Dynamic Splinting Increases Flexion for Hallux Rigidus. BioMechanics, 2007 Sept;14(9), pg49-53
- [Background] Willis B. Post-TBI Gait Rehabilitation. Applied Neurol. 2007 Jul;3(7):25-26
- [Background] Lemont H, Ammirati KM, Usen N. Plantar fasciitis: a degenerative process (fasciosis) without inflammation. J Am Podiatr Med Assoc. 2003 May-Jun;93(3):234-7. doi: 10.7547/87507315-93-3-234. PMID 12756315
- [Background] Martin JE, Hosch JC, Goforth WP, Murff RT, Lynch DM, Odom RD. Mechanical treatment of plantar fasciitis. A prospective study. J Am Podiatr Med Assoc. 2001 Feb;91(2):55-62. doi: 10.7547/87507315-91-2-55. PMID 11266478
- [Background] Ng A, Beegle T, Rockett AK. Atypical presentation of plantar fasciitis secondary to soft-tissue mass infiltration. J Am Podiatr Med Assoc. 2001 Feb;91(2):89-92. doi: 10.7547/87507315-91-2-89. PMID 11266484
- [Background] Hart LE. Exercise and soft tissue injury. Baillieres Clin Rheumatol. 1994 Feb;8(1):137-48. doi: 10.1016/s0950-3579(05)80228-6. PMID 8149440
- [Background] Intenzo CM, Wapner KL, Park CH, Kim SM. Evaluation of plantar fasciitis by three-phase bone scintigraphy. Clin Nucl Med. 1991 May;16(5):325-8. doi: 10.1097/00003072-199105000-00006. PMID 2054987
- [Background] Hepburn, G. Contracture and Stiff Joint Management with Dynasplint®. J Ortho Sports Phys Ther. 1987;8(10): 498-504
- See also: Related Info — http://www.dynasplint.com